CLINICAL TRIAL: NCT00910208
Title: Safety and Efficacy of Patient Controlled Analgesia in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH); Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-448; 1R21NR010929-01 (NIH)
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Pain
Keywords: Pain; Analgesia; Analgesia, Patient-controlled; Emergency Medicine
MeSH Terms: conditions — Pain; Agnosia | interventions — Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patient-controlled analgesia 1 mg demand dose (Experimental): 0.1 mg/kg morphine loading dose plus PCA with 1.0 mg morphine demand dosing every 6 minutes
  Interventions: Device: Patient-controlled analgesia; Drug: morphine
- Patient-controlled analgesia 1.5 mg demand dose (Experimental): 0.1 mg/kg morphine loading dose plus PCA with 1.5 mg morphine demand dosing every 6 minutes
  Interventions: Device: Patient-controlled analgesia; Drug: morphine
- Non-Patient-controlled analgesia comparison group (Active Comparator): 0.1 mg/kg morphine loading dose plus additional analgesia as needed
  Interventions: Drug: morphine

INTERVENTIONS:
Device: Patient-controlled analgesia — Intravenous morphine delivered via Curlin painsmart PCA device
  Other Names: PCA
  Arms: Patient-controlled analgesia 1 mg demand dose; Patient-controlled analgesia 1.5 mg demand dose
Drug: morphine — Intravenous morphine

SUMMARY:
The aims of this study are to assess efficacy and safety of patient-controlled analgesia (PCA) when applied to the Emergency Department setting and to compare the efficacy and safety of two PCA dosing regimens.

DETAILED DESCRIPTION:
The safety, efficacy, and dosing of PCA will be assessed in a randomized trial with three treatment arms:

1. PCA with 1.0 mg morphine demand dosing every 6 minutes,
2. PCA with 1.5 mg demand dosing every 6 minutes and
3. a non-PCA comparison group.

All patients will receive a loading dose of 0.1 mg/kg morphine. All patients can receive additional analgesics as needed, at the discretion of the provider.

We hypothesize that morphine supplied via PCA will provide superior analgesia without a greater incidence of adverse events when compared to non-PCA pain management; and that PCA demand dosing of 1.5 mg will be superior to 1.0 mg without more adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the ED with a chief complaint of abdominal pain of less than or equal to 7 days duration
* Age 18 to 65 years
* Patient deemed by the ED attending physician to require IV opioid analgesia

Exclusion Criteria:

* Current use of prescription or non-prescription opioids
* Long-term use of opioids, chronic pain syndrome
* Clinician suspicion of opioid dependence/abuse
* Clinical suspicion of intoxication
* Pregnancy or breast-feeding
* History of chronic obstructive pulmonary disease, history of sleep apnea, oxygen saturation < 97%
* Systolic blood pressure < 100 mm Hg
* Use of monoamine oxidase inhibitors, phenothiazines, or tricyclic antidepressants
* History of renal insufficiency/renal failure
* Prior allergic reaction to morphine
* Inability to provide informed consent
* Previous entry of patient into study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne J Birnbaum, MD, MS, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine; Polly E Bijur, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Birnbaum A, Schechter C, Tufaro V, Touger R, Gallagher EJ, Bijur P. Efficacy of patient-controlled analgesia for patients with acute abdominal pain in the emergency department: a randomized trial. Acad Emerg Med. 2012 Apr;19(4):370-7. doi: 10.1111/j.1553-2712.2012.01322.x. PMID 22506940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started April 3, 2009 and ended June 30, 2010. Patients were recruited by bilingual research associates in the Emergency Department of Jacobi Medical Center, Bronx, NY
Groups:
- PCA 1 mg Demand Dose: 0.1 mg/kg morphine loading dose followed by PCA with 1.0 mg morphine demand dose every 6 minutes
  Patient-controlled analgesia: Intravenous morphine delivered via Curlin painsmart PCA device
  morphine: Intravenous morphine
- PCA 1.5 mg Demand Dose: 0.1 mg/kg morphine loading dose followed by PCA with 1.5 mg morphine demand dosing every 6 minutes
  Patient-controlled analgesia: Intravenous morphine delivered via Curlin painsmart PCA device
  morphine: Intravenous morphine
- Non-PCA Comparison Group: 0.1 mg/kg morphine loading dose followed by additional analgesia supplemented as needed at the discretion of the treating physician, using usual procedures for monitoring and treating pain.
  morphine: Intravenous morphine
Period: Overall Study
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Started | 69 | 72 | 70
Completed | 67 | 70 | 69
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- PCA 1 mg Demand Dose: 0.1 mg/kg morphine loading dose followed by PCA with 1.0 mg morphine demand dosing every 6 minutes
  Patient-controlled analgesia: Intravenous morphine delivered via Curlin painsmart PCA device
  morphine: Intravenous morphine
- Total: Total of all reporting groups
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group | Total
Number analyzed (Participants) | 67 | 70 | 69 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10) | 38 (12) | 37 (12) | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 47 | 51 | 141
  Male | 24 | 23 | 18 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnicity were asked separately. As the majority of patients who identified their ethnicity as Hispanic/Latino did not specify a race, patients were categorized as Hispanic/Latino regardless of race. If patients were not Hispanic/Latino, they were categorized by race
  Participants
    Hispanic/Latino | 41 | 46 | 37 | 124
    Black/African American - not Hispanic | 16 | 15 | 25 | 56
    White - not Hispanic | 3 | 4 | 5 | 12
    Asian/other | 7 | 5 | 2 | 14
Initial Pain Score [Count of Participants; unit: Participants] — Numerical rating scale (NRS) of pain: 0 indicates no pain, 10 indicates worst possible pain
  Participants
    Pain Score less than 7 | 6 | 4 | 4 | 14
    Pain Score=7 | 5 | 6 | 13 | 24
    Pain Score=8 | 8 | 17 | 10 | 35
    Pain Score=9 | 11 | 11 | 11 | 33
    Pain Score=10 | 37 | 32 | 31 | 100

OUTCOME MEASURES:

1. Primary Outcome: Short Term Efficacy: Change in Pain Intensity as Assessed by Patient Self Report on Numerical Rating Scale
Description: Participants will complete a survey in which they rate their pain on a Numerical Rating Scale (NRS) of pain ranging from 0 - no pain, to 10 - worst imaginable pain, higher scores indicate worse pain. Change is measured by subtracting the 30 minute NRS score from the Baseline NRS score, thus higher numbers indicate greater decrease in pain, negative numbers indicate increase in pain from baseline to 30 minutes post-baseline.
Time Frame: Baseline and 30 minutes post treatment
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Number analyzed (Participants) | 67 | 70 | 69
Units on a scale | 3.8 [3.0 to 4.6] | 4.0 [3.3 to 4.6] | 3.6 [2.9 to 4.4]
Statistical Analysis 1: Comparison: PCA 1 mg Demand Dose vs PCA 1.5 mg Demand Dose vs Non-PCA Comparison Group; Test type: Superiority; p = 0.82, ANOVA

2. Primary Outcome: Participants With Short Term Efficacy: Pain Relief by 30 Minutes
Description: Pain Intensity measured on Likert Scale. Participants self report pain level according to the scale by selecting from No relief, Slight relief, Moderate relief, A lot of relief, and Complete relief)
Time Frame: 30 minutes post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Number analyzed (Participants) | 67 | 70 | 69
Participants
  No relief | 4 | 4 | 4
  Slight relief | 14 | 10 | 16
  Moderate relief | 18 | 20 | 12
  A lot of relief | 24 | 31 | 25
  Complete relief | 7 | 5 | 12
Statistical Analysis 1: Comparison: PCA 1 mg Demand Dose vs PCA 1.5 mg Demand Dose vs Non-PCA Comparison Group; Test type: Superiority; p = 0.47, Chi-squared

3. Primary Outcome: Long Term Efficacy: Total Analgesia Provided Over 2 Hours
Description: Participants will complete a survey in which they rate their pain on a Numerical Rating Scale (NRS) of pain ranging from 0 - no pain, to 10 - worst imaginable pain, higher scores indicate worse pain
  Total analgesia is measured by a summary of change in pain that varies from 0 - no change to
Time Frame: Baseline, 30, 60, 90, 120 post-treatment
Measure: Mean (95% Confidence Interval); unit: scores on a scale *minutes
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Number analyzed (Participants) | 67 | 70 | 69
scores on a scale *minutes | -16.4 [-18.8 to -14.1] | -17.4 [-19.7 to -15.1] | -13.6 [-15.9 to -11.3]
Statistical Analysis 1: Comparison: PCA 1 mg Demand Dose vs PCA 1.5 mg Demand Dose vs Non-PCA Comparison Group; Test type: Superiority; p = 0.06, ANOVA

4. Primary Outcome: Long Term Efficacy: Pain Relief by 120 Minutes
Description: Participants aksed to and give range
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Number analyzed (Participants) | 65 | 69 | 68
Participants
  No relief | 7 | 6 | 6
  Slight relief | 9 | 5 | 18
  Moderate relief | 9 | 8 | 13
  A lot of relief | 22 | 34 | 16
  Complete relief | 18 | 16 | 15
Statistical Analysis 1: Comparison: PCA 1 mg Demand Dose vs PCA 1.5 mg Demand Dose vs Non-PCA Comparison Group; Test type: Superiority; p = 0.033, Chi-squared

5. Primary Outcome: Safety: Incidence of Adverse Events
Description: Adverse Events defined as: oxygen saturation < 92%; respiratory rate <10 breaths/min; systolic blood pressure < 90 mm Hg)
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Number analyzed (Participants) | 67 | 70 | 69
Participants
  1 or more adverse events | 0 | 1 | 1
  No Adverse events | 67 | 69 | 68
Statistical Analysis 1: Comparison: PCA 1 mg Demand Dose vs PCA 1.5 mg Demand Dose vs Non-PCA Comparison Group; Test type: Superiority; p = 0.99, Fisher Exact

6. Secondary Outcome: Need for Supplementary Analgesia
Description: count of participants who needed or did not needed additional analgesia
Time Frame: 2 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
Number analyzed (Participants) | 67 | 70 | 69
Participants
  Needed supplementary medication | 4 | 0 | 20
  Did not need supplementary medication | 63 | 70 | 49
Statistical Analysis 1: Comparison: PCA 1 mg Demand Dose vs PCA 1.5 mg Demand Dose vs Non-PCA Comparison Group; Test type: Superiority; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 8 hours
Arm/Group | PCA 1 mg Demand Dose | PCA 1.5 mg Demand Dose | Non-PCA Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/70 | 1/69
Other Adverse Events (participants affected / at risk) | 1/67 | 0/70 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCA 1 mg Demand Dose (N=67) | PCA 1.5 mg Demand Dose (N=70) | Non-PCA Comparison Group (N=69)
Transient Oxygen Desaturation as measured by pulse oximetry (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Transient decrease in blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCA 1 mg Demand Dose (N=67) | PCA 1.5 mg Demand Dose (N=70) | Non-PCA Comparison Group (N=69)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Transient sluggish response to loud sound after also receiving lorazepam (non-study drug)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No